CLINICAL TRIAL: NCT05181306
Title: Long-term Oncologic Outcomes of Robotic Versus Laparoscopic Total Gastrectomy for Advanced Gastric Cancer: A Propensity Score Matching Study
Brief Title: Long-term Oncologic Outcomes of Robotic Versus Laparoscopic Total Gastrectomy for Advanced Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Yan Shi, Head of General Surgery, Southwest Hospital, China
Other Study IDs: KY2021123
Record Dates: First submitted 2021-12-06; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Gastric Cancer
Keywords: Advanced gastric cancer; Total gastrectomy; Robotic; Laparoscopic; Long-term outcomes
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robotic surgery
  Interventions: Procedure: Robotic-assisted Total Gastrectomy with D2 Lymphadenectomy
- Laparoscopic surgery
  Interventions: Procedure: Laparoscopic-assisted Total Gastrectomy with D2 Lymphadenectomy

INTERVENTIONS:
Procedure: Robotic-assisted Total Gastrectomy with D2 Lymphadenectomy — Robotic-assisted total gastrectomy with D2 lymph node dissection will be performed with curative treated intent according to the patients' or their legal representatives'willing to choose robotic-assisted total gastrectomy and excluding T4b、bulky lymph nodes or distant metastasis case by diagnostic laparoscopy. The alimentary canal reconstruction method is selected as esophageal jejunal R-Y anastomosis. Whether to reinforce the anastomotic manually is decided by the surgeon's experience. The reconstruction can be carried out by extracorporeal or intracorporeal anastomosis.
  Groups: Robotic surgery
Procedure: Laparoscopic-assisted Total Gastrectomy with D2 Lymphadenectomy — Laparoscopic-assisted total gastrectomy with D2 lymph node dissection will be performed with curative treated intent according to the patients' or their legal representatives'willing to choose laparoscopic-assisted total gastrectomy and excluding T4b、bulky lymph nodes or distant metastasis case by diagnostic laparoscopy. The alimentary canal reconstruction method is selected as esophageal jejunal R-Y anastomosis. Whether to reinforce the anastomotic manually is decided by the surgeon's experience. The reconstruction can be carried out by extracorporeal or intracorporeal anastomosis.
  Groups: Laparoscopic surgery

SUMMARY:
This study is a retrospective, single-center, controlled and observation trial comparing robotic total gastrectomy with D2 lymph nodal dissection for locally advanced gastric cancer patients with laparoscopic procedure.

DETAILED DESCRIPTION:
Since Kitano firstly reported laparoscopy-assisted distal gastrectomy in 1994, the number of patients undergoing the laparoscopic procedure has gradually increased. The latest Japanese gastric cancer treatment guideline recommends laparoscopic gastrectomy (LG) as an optional treatment for cStage（clinical stage） Ⅰ gastric cancer (GC).

Based on the experience of early GC, most experienced surgeons have applied the laparoscopic procedure in patients with locally advanced gastric cancer (AGC) especially in east world like China, Japan and Korea. Though applying laparoscopic total gastrectomy (LTG) is much more difficulty than that of distal gastrectomy (DG), there are a mount of centers reported their experiences of this procedure. A meta-analysis including seventeen studies of 2313 patients (955 in LTG and 1358 in open total gastrectomy) demonstrated that LTG can have less blood loss, fewer analgesic uses, earlier passage of flatus, quicker resumption of oral intake, earlier hospital discharge, and reduced postoperative morbidity. However, the number of harvested lymph nodes, proximal resection margin, hospital mortality, 5-year OS(overall survival) and DFS(disease-free survival) were similar in both groups. According to the existing reports, LTG is technically safety and feasibility.

To overcome the limitations of laparoscopic surgery, robot systems have been introduced to treat GC providing technical advantages since Hashizume firstly reported. Yoon and Son respectively compared robot total gastrectomy (RTG) with LTG, they drew a common conclusion that the number of dissected lymph nodes and postoperative complications were similar in both groups. But Son found that the mean numbers of retrieved lymph nodes along the splenic artery from RTG was higher than LTG (2.3 vs. 1.0, p = 0.013), as was also the case at the splenic hilum and artery (3.6 vs.1.9, p = 0.014). Regretfully, most of their reported cases were early gastric cancer (EGC). Other literatures reported AGC patients under RTG or LTG together with distal gastrectomy (DG), the investigators haven't found any literature compare RTG with LTG alone for AGC retrospectively.

Since most literatures are EGC patients and retrospectively researches, the investigators can't insist that patients with AGC may benefit under RTG. Therefore, the investigators launch this retrospective, single-center, controlled observation trial comparing RTG for locally advanced gastric cancer patients with LTG. In the process of research, it will be divided into two groups according to the willing of patients or their legal representatives who choose one of the two procedures(RTG or LTG) to cure GC.

ELIGIBILITY:
Inclusion Criteria:

* 1.Pathologically proven gastric adenocarcinoma; 2.Age: older than 18 years old, younger than 80 years old; 3.Tumor located in the upper third of the stomach or esophagogastric junction or other location, and is possible to be curatively resected by total gastrectomy; 4.Preoperative stage of cT2-4aN0-3M0 according to American Joint Committee on Cancer/Union for International Cancer Control 8th edition; 5.American Society of Anesthesiology (ASA) score of class I to III; 6.Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; 7.Patients who freely give informed consent to participate in the clinical study;

Exclusion Criteria:

* 1.Early gastric cancer; 2.Age: younger than 18 years old, older than 80 years old; 3.Total gastrectomy with D2 lymphadenectomy was not required; 4.Enlarged or bulky regional lymph node diameter larger than 3 cm based on preoperative imaging; 5.Emergency surgery for gastric cancer-related complications (bleeding or complete obstruction or perforation); 6.Previous upper abdominal surgery (except laparoscopic cholecystectomy); 7.Previous neoadjuvant chemotherapy or radiotherapy for gastric cancer; 8.Unstable angina or myocardial infarction within the past 6 months; 9.Cerebrovascular accident within the past 6 months; 10.American Society of Anesthesiology (ASA) score of class more than III; 11.Severe respiratory disease (FEV1< 50%); 12.Continuous systemic steroid therapy within 1 month before the study; 13.Pregnant or breast-feeding women;

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with gastric cancer who need to received total gastrectomy with D2 lymphadenectomy.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
5-year Overall survival rate | 5 years
  5-year Overall survival rate
5-year Disease-free survival rate | 5 years
  5-year Disease-free survival rate
Recurrence | 5 years
  Recurrence

SECONDARY OUTCOMES:
Overall postoperative morbidity and mortality | 30 days
  Refers to the incidence of early postoperative complications. The early postoperative complication are defined as the event observed within 30 days after surgery.
Time of operation | 1 day
  The total time of operation
Estimated blood loss | 1 day
  Blood loss during intraoperative including the volume of negative pressure drainage bottle and the increasing weight of gauzes （ml）
Blood transfusion | 1 day
  Blood transfusion during operation
Length of proximal and distal cutting margin | 1 day
  Length of proximal and distal cutting margin of the specimen
Number of retrieved overall lymph nodes, N1 lymph nodes, N2 lymph nodes and supra-pancreatic lymph nodes | 7 days
  Number of retrieved overall lymph nodes, N1 lymph nodes, N2 lymph nodes and supra-pancreatic lymph nodes
Time to flatus | 30 days
  Time of anus exsufflation
Time to liquid diet | 30 days
  Time to liquid diet
Time to soft diet | 30 days
  Time to soft diet
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay
Cost | 30 days
  All costs of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Pei-wu Yu, Study Chair — Department of General Surgery and Center of Microinvasive Gastrointestinal Surgery,Southwest Hospital
Locations (1):
- Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2014 (ver. 4). Gastric Cancer. 2017 Jan;20(1):1-19. doi: 10.1007/s10120-016-0622-4. Epub 2016 Jun 24. No abstract available. PMID 27342689
- [Background] Etoh T, Honda M, Kumamaru H, Miyata H, Yoshida K, Kodera Y, Kakeji Y, Inomata M, Konno H, Seto Y, Kitano S, Hiki N. Morbidity and mortality from a propensity score-matched, prospective cohort study of laparoscopic versus open total gastrectomy for gastric cancer: data from a nationwide web-based database. Surg Endosc. 2018 Jun;32(6):2766-2773. doi: 10.1007/s00464-017-5976-0. Epub 2017 Dec 7. PMID 29218676
- [Background] Yoon HM, Kim YW, Lee JH, Ryu KW, Eom BW, Park JY, Choi IJ, Kim CG, Lee JY, Cho SJ, Rho JY. Robot-assisted total gastrectomy is comparable with laparoscopically assisted total gastrectomy for early gastric cancer. Surg Endosc. 2012 May;26(5):1377-81. doi: 10.1007/s00464-011-2043-0. Epub 2011 Nov 16. PMID 22083338
- [Background] Son T, Lee JH, Kim YM, Kim HI, Noh SH, Hyung WJ. Robotic spleen-preserving total gastrectomy for gastric cancer: comparison with conventional laparoscopic procedure. Surg Endosc. 2014 Sep;28(9):2606-15. doi: 10.1007/s00464-014-3511-0. Epub 2014 Apr 3. PMID 24695982
- [Background] Shen W, Xi H, Wei B, Cui J, Bian S, Zhang K, Wang N, Huang X, Chen L. Robotic versus laparoscopic gastrectomy for gastric cancer: comparison of short-term surgical outcomes. Surg Endosc. 2016 Feb;30(2):574-580. doi: 10.1007/s00464-015-4241-7. Epub 2015 Jul 25. PMID 26208497
- [Background] Pan HF, Wang G, Liu J, Liu XX, Zhao K, Tang XF, Jiang ZW. Robotic Versus Laparoscopic Gastrectomy for Locally Advanced Gastric Cancer. Surg Laparosc Endosc Percutan Tech. 2017 Dec;27(6):428-433. doi: 10.1097/SLE.0000000000000469. PMID 29211699
- [Background] Junfeng Z, Yan S, Bo T, Yingxue H, Dongzhu Z, Yongliang Z, Feng Q, Peiwu Y. Robotic gastrectomy versus laparoscopic gastrectomy for gastric cancer: comparison of surgical performance and short-term outcomes. Surg Endosc. 2014 Jun;28(6):1779-87. doi: 10.1007/s00464-013-3385-6. Epub 2014 Jan 3. PMID 24385251
- [Background] Wang W, Zhang X, Shen C, Zhi X, Wang B, Xu Z. Laparoscopic versus open total gastrectomy for gastric cancer: an updated meta-analysis. PLoS One. 2014 Feb 18;9(2):e88753. doi: 10.1371/journal.pone.0088753. eCollection 2014. PMID 24558421